CLINICAL TRIAL: NCT06070246
Title: Gaining Insights Into Patient Involvement Patterns and Trends in Participation in Lymphoma Clinical Trials
Brief Title: Navigating the Clinical Research Process for Lymphoma
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 71918699
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Lymphoma
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in medical research usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This trial will admit a wide range of data on the clinical trial experience of lymphoma patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of lymphoma
* Participant must be 18 years of age or older
* Participant must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study.

Exclusion Criteria:

* Pregnant or lactating woman
* Participant is actively receiving study therapy in another
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lymphoma patients who are actively considering participating in a clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a lymphoma clinical research. | 3 months
Number of lymphoma study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He X, Xu P, Wang X, Jiang S, Gong D, Wu N. The association of gene rearrangement and lymphoma diagnosis: A prospective observational study. Medicine (Baltimore). 2020 Jun 12;99(24):e20733. doi: 10.1097/MD.0000000000020733. PMID 32541525
- [Background] Dhir V, Maganti M, Rozenberg D, Kukreti V, Kuruvilla J, Crump M, Prica A. Predicting the Risks of Aggressive-Intent Chemotherapy Toxicity in Older Patients With Lymphoma: A Prospective Observational Pilot Study. Clin Lymphoma Myeloma Leuk. 2022 Aug;22(8):e792-e803. doi: 10.1016/j.clml.2022.04.011. Epub 2022 Apr 29. PMID 35650009
- [Background] Tanaka R, Kaburaki T, Taoka K, Karakawa A, Tsuji H, Nishikawa M, Yatomi Y, Shinozaki-Ushiku A, Ushiku T, Araki F. More Accurate Diagnosis of Vitreoretinal Lymphoma Using a Combination of Diagnostic Test Results: A Prospective Observational Study. Ocul Immunol Inflamm. 2022 Aug;30(6):1354-1360. doi: 10.1080/09273948.2021.1873394. Epub 2021 Apr 1. PMID 33793360

DOCUMENTS (1):
  • Informed Consent Form (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT06070246/ICF_000.pdf